CLINICAL TRIAL: NCT04194008
Title: An Open Label, Single Arm, Multicenter Study Assessing the Efficacy and Safety of Nerivio, a Remote Electrical Neuromodulation Device, for Acute Treatment of Migraine in People With Chronic Migraine
Brief Title: Efficacy and Safety of Nerivio Device for Acute Treatment of Migraine in People With Chronic Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theranica (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TCH006
Record Dates: First submitted 2019-12-04; First posted 2019-12-11 (Actual); Results first posted 2021-02-02 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2020-09

CONDITIONS: Chronic Migraine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Nerivio device treatment (Experimental): Treatment with active Nerivio device
  Interventions: Device: Nerivio

INTERVENTIONS:
Device: Nerivio — A remote electrical neuromodulation (REN) device for the acute treatment of migraines.The device delivers transcutaneous electrical stimulation to the upper arm to induce conditioned pain modulation (CPM) that activates a descending endogenous analgesic mechanism. The treatment is self-administered and controlled by a smartphone application.

SUMMARY:
A prospective, single arm, open-label, multicenter trial to assess the efficacy and safety of the Nerivio device in chronic migraine patients. This study will be conducted in three phases:

Phase I - Run-in:

Eligible participants will be trained to use a smartphone migraine diary application. During the 4 weeks of this phase, participants will be instructed to report all their migraines and headaches at onset, 2 hours and 24 hours post report .

Phase II - Treatment:

A 4-week treatment phase in which participants will be asked to treat their migraine headaches with the Nerivio device and report it using the smartphone application at baseline, 2 hours and 24 hours post-treatment.

Phase III - Follow-up:

An 8-week follow-up phase in which participants will incorporate the Nerivio device into their usual care according to their preference (Nerivio only, medication only, both or none). Participants will be asked to report all their migraines or headaches at onset, 2 hours post report and 24 hours post report.

DETAILED DESCRIPTION:
This open label study includes up to four visits. The enrollment and application training may occur in two separate visits instead of one.

First visit - The first visit will include screening, enrollment and training on the application.

Enrollment: The screening process will include an eligibility assessment and a urine pregnancy test. Following successful screening, the site staff will provide the participants with study related information, perform an enrollment interview and receive an informed consent from the participants. During this visit, participants will complete baseline questionnaires that included information on the frequency and severity of their migraine attacks, typical associated symptoms, use of preventive and acute treatments, and the effect that their migraine attacks have on their daily routine and quality of life.

Application training: Eligible participants who enroll to the study will be trained to use the diary mode of the application that is installed on their own smartphones. The participants will be instructed to report the onset of all their migraines and headaches and complete a migraine diary questions regarding their pain intensity levels, the presence/absence of aura and associated migraine symptoms (nausea, photophobia, phonophobia, and allodynia) as well as rate their stress level and functional disability at baseline, 2- and 24-hours post-treatment. At the beginning of each treatment, participants will also be asked to report the time elapsed from attack onset. The site personnel will be required to document the training session in the Case Report Form (CRF).

Run-in phase: After the enrollment visit, participants will undergo a 4-week migraine diary phase aimed to collect baseline migraine characteristics and further assess eligibility. The participants will use the app to record pain intensity levels, the presence/absence of aura and associated migraine symptoms (nausea, photophobia, phonophobia, and allodynia) as well as the effect that their migraine attacks have on their daily routine and quality of life, at baseline, 2- and 24-hours post-treatment. These reports will be transferred by the application to the electronic data capture (EDC) system, where they will be collected and registered.

Participants who report at least 6 qualifying migraine headaches with pain data at baseline and 2 hours post-treatment will continue to the treatment phase.

Second visit- Device training: Eligible participants who successfully complete the run-in phase will receive the Nerivio™ device. The device will be registered and connected by Bluetooth to their smartphone. During this visit, participants will be trained to use the device. Device training will include finding the optimal individual stimulation intensity level (perceptible but not painful), that will be subject to change during the treatment phase. The site staff will also carefully review with the patient how to identify a qualifying migraine headache (see below) and provide detailed instructions on study procedures.

If the research staff recognizes that the participant cannot tolerate the feeling of the electrical stimulation, the participant may be withdrawn from the study.

During the training, participants will also be informed on the key elements which are critical for the successful conduct of the study:

* Treatments of migraine and headaches with Nerivio™ should be performed as soon as possible after migraine headache or aura began and always within one hour of symptoms onset. Treatments of mild headaches are accepted.
* Avoid taking rescue medications within two hours post-treatment (2 hours from start of treatment), if possible.
* The treatment should be performed for at least 30 minutes (the recommended treatment duration is 45 minutes).

The site personnel will be required to document the training session in the CRF.

Treatment phase: Participants will be instructed to use the device for the treatment of migraine and/or headaches (see below) as soon as possible and always within 60 minutes of onset during a period of up to 4 weeks. Participants will be instructed to use the device with the intensity level identified during the device training visit (and adjust as necessary) and make sure the stimulation is perceptible but not painful. Participants will be instructed to avoid taking rescue medications within 2 hours post-treatment. If medications are used, participants will be instructed to record in the app when and which medication was taken at 2- and 24-hours post treatment. The participants will use the app to record pain intensity levels, the presence/absence of aura and associated migraine symptoms (nausea, photophobia, phonophobia, and allodynia) as well as the effect that their migraine attacks have on their daily routine and quality of life, at baseline, 2- and 24-hours post-treatment. At the beginning of each treatment, participants will also be asked to report the time elapsed from attack onset. Adverse events will be reported throughout this phase of the study directly to the site staff.

Participants who do not achieve satisfactory relief at 2 hours post-treatment may treat again with the Nerivio™ device or may treat with usual care at that time or any time thereafter if the headache does not resolve. Participants will also be able to treat headache recurrence with the device. Migraine headaches that are not treated with the device may be treated with usual care.

The first reported treatment will be considered a "training" treatment, aimed to verify that the participants use the device properly, and will only be included in the safety analysis. The efficacy evaluation will be performed on the first treatment of a qualifying attack (see below) following the training treatment (hereby termed "test treatment").

Third visit- Follow-up phase:

Following the 4-week period of the treatment phase, participants will return to the clinic to fill questionnaires assessing satisfaction and user experience. All participants who complete the treatment phase will enter an additional 8-week phase in which the device can be incorporate into their usual care. Participants will treat their migraines and headaches according to their preference- treatment with Nerivio only, treatment with medication only, both treatment options, or none. Participants will be asked to report all their migraine headaches at onset (migraines or headache), regardless if they are using the device or not. The participants will use the app to record pain intensity levels, the presence/absence of aura and associated migraine symptoms (nausea, photophobia, phonophobia, and allodynia) as well as the effect that their migraine attacks have on their daily routine and quality of life, at baseline, 2- and 24-hours post-treatment.

Fourth (final) visit - End of study:

Participants will return to the clinic following the end of the follow-up phase, at which time they will return the device. The participants will have the option of returning the device by mail instead of an on-site visit. Participants may be asked to fill additional questionnaires on their migraine and their experience with the device.

ELIGIBILITY:
Inclusion Criteria:

1. Participants aged 18-75 years old.
2. Participants meeting the International Classification of Headache Disorders-3 (ICHD-3) diagnostic criteria for chronic migraine
3. Participants experiencing between 15 to 23 headache days per month, with at least 8 headache days (per month) with migraine phenotype presentation
4. Participants have personal access to a smartphone
5. Participants must be able and willing to comply with the protocol
6. Participants must be able and willing to provide written informed consent

Exclusion Criteria:

1. Participants with an active implanted electrical and/or neurostimulator device (e.g. cardiac pacemaker, cochlear implant).
2. Participants with congestive heart failure (CHF), severe cardiac or cerebrovascular disease.
3. Participants with uncontrolled epilepsy.
4. Lack of efficacy, after an adequate therapeutic trial, of at least two migraine specific acute medications.
5. Change in migraine preventive medications (type or dose) in the last two months prior to recruitment and/or during the study
6. Pregnant, trying to get pregnant or breastfeeding female participants
7. Subjects participating in any other interventional clinical study.
8. Participants without basic cognitive and/or motor skills needed to operate a smartphone
9. Participants with other significant pain, medical or psychological problems that in the opinion of the investigator may confound the study assessments
10. Participants who have previous experience with the device

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-11-18 (Actual); Primary Completion 2020-05-22 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Grosberg, MD, Principal Investigator — Hartford Healthcare Center
Locations (10):
- United States (10):
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - California Medical Clinic for Headache, Santa Monica, California
  - Hartford Healthcare Center, Hartford, Connecticut
  - Headache Neurology Research Institute, Ridgeland, Mississippi
  - StudyMetrix Research, LLC, City of Saint Peters, Missouri
  - ClinVest, Springfield, Missouri
  - Mercy Hospital, St Louis, Missouri
  - Island Neurological, Plainview, New York
  - Preferred Primary Care Physicians, Inc., Pittsburgh, Pennsylvania
  - Nashville neuroscience, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grosberg B, Rabany L, Lin T, Harris D, Vizel M, Ironi A, O'Carroll CP, Schim J. Safety and efficacy of remote electrical neuromodulation for the acute treatment of chronic migraine: an open-label study. Pain Rep. 2021 Oct 14;6(4):e966. doi: 10.1097/PR9.0000000000000966. eCollection 2021 Nov-Dec. PMID 34667919

RESULTS

PARTICIPANT FLOW:
Period: Baseline (Run-in) Phase
Arm/Group | Nerivio Device Treatment
Started | 126
Completed | 99
Not Completed | 27
Not completed — Fail to comply with Run-in phase criteria | 19
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 2
Period: Treatment Phase With Nerivio
Arm/Group | Nerivio Device Treatment
Started | 99
Completed | 91
Not Completed | 8
Not completed — Withdrawal by Subject | 3
Not completed — Missing data | 4
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 126
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 110
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 115
  More than one race | 0
  Unknown or Not Reported | 3
Average number of headache days per month [Mean (Standard Deviation); unit: Days] | 18.8 (2.7)
Average number of migraine headache days per month [Mean (Standard Deviation); unit: Days] | 16.4 (3.7)
Use of preventive medication [Count of Participants; unit: Participants] | 80
Migraine with aura [Count of Participants; unit: Participants] | 36
Triptan usage [Count of Participants; unit: Participants] | 49

OUTCOME MEASURES:

1. Primary Outcome: Pain Relief at 2 Hours Post-treatment
Description: The proportion of subjects reporting, for the test treatment, pain relief at 2 hours post-treatment without the use of rescue medication. Pain relief is defined as an improvement from severe or moderate pain to mild or no pain, or from mild pain to no pain. Pain level will be reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain, 3- Severe pain)
Time Frame: 2 hours post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 91
Participants | 54

2. Secondary Outcome: Pain-free at 2 Hours Post-treatment
Description: The proportion of subjects reporting, for the test treatment, no pain at 2 hours post-treatment without the use of rescue medication. Pain-free is defined as improvement from mild, moderate, or severe pain to none. Pain level will be reported using a 4-point Likert scale (0 - No pain, 1 - Mild pain, 2 - Moderate pain, 3- Severe pain)
Time Frame: 2 hours post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 91
Participants | 19

3. Secondary Outcome: Disappearance of Nausea at 2 Hours Post-treatment
Description: The proportion of subjects presented nausea at the migraine onset and reported disappearance of nausea at 2 hours post-treatment of the test treatment
Time Frame: 2 hours post treatment
Population: only 41 participants reported nausea at T=0 hours. thus, this is the denominator number for this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 41
Participants | 20

4. Secondary Outcome: Disappearance of Photophobia at 2 Hours Post-treatment
Description: The proportion of subjects presented photohobia at the migraine onset and reported disappearance of photophobia at 2 hours post-treatment of the test treatment
Time Frame: 2 hours post treatment
Population: only 74 participants reported photophobia at T=0 hours. thus, this is the denominator number for this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 74
Participants | 30

5. Secondary Outcome: Disappearance of Phonophobia at 2 Hours Post-treatment
Description: The proportion of subjects presented phonophobia at the migraine onset and reported disappearance of phonophobia at 2 hours post-treatment of the test treatment
Time Frame: 2 hours post treatment
Population: only 65 participants reported phonophobia at T=0 hours. thus, this is the denominator number for this analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 65
Participants | 29

6. Other Pre Specified Outcome: Within-subject Consistency of the Pain Relief Response
Description: proportion of patients achieving pain relief at 2 hours in at least 50% of all their treatments
Time Frame: throughout the study
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 91
Participants | 52

7. Other Pre Specified Outcome: Functional Disability at 2 Hours Post-treatment
Description: The proportion of participants achieving improvement of at least one grade in functional disability in the test treatment at 2 hours post-treatment with no use of rescue medication
Time Frame: 2 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 32
Participants | 19

8. Other Pre Specified Outcome: Functional Disability at 24 Hours Post-treatment
Description: The proportion of participants achieving improvement of at least one grade in functional disability in the test treatment at 24 hours post-treatment with no use of rescue medication
Time Frame: 24 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 14
Participants | 7

9. Other Pre Specified Outcome: Sustained Pain Relief at 24 Hours Post-treatment
Description: The proportion of subjects achieving, for the test treatment, pain relief at 2 hours post-treatment without the use of rescue medication and no relapse of headache pain within 24 hours
Time Frame: 24 hours post treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Nerivio Device Treatment
Number analyzed (Participants) | 45
Participants | 33

ADVERSE EVENTS:
Time Frame: Up to 12 weeks
Description: The Nerivio device is a neurostimulator and it is externally applied over the body. The Nerivio is accepted as a non-significant risk (NSR) device. In addition, as the exclusion criteria for the study leave out participant with electrical implant, congenital heart failure or epilepsy, the number of high risk participants is zero.
Arm/Group | Nerivio Device Treatment
All-Cause Mortality (participants affected / at risk) | 0/99
Serious Adverse Events (participants affected / at risk) | 0/99
Other Adverse Events (participants affected / at risk) | 9/99
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nerivio Device Treatment (N=99)
Pain in the arm (Nervous system disorders) | 1 (1)
Sinus infection (Infections and infestations) | 1 (1)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Ear infection (Infections and infestations) | 1 (1)
viral infectioniral infection (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Leg pain (Nervous system disorders) | 1 (1)
Poison ivy rash (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
No limitations or caveats were reported

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04194008/Prot_SAP_000.pdf
  • Informed Consent Form (2019-09-01): https://cdn.clinicaltrials.gov/large-docs/08/NCT04194008/ICF_001.pdf